CLINICAL TRIAL: NCT02850861
Title: A New Surgical Instrument in Treatment of Conlylar Fracture: Condylar Reductor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Junhui Cui (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor-Investigator, Junhui Cui, Principal investigator, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: WCH-01
Record Dates: First submitted 2016-07-06; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Mandibular Fracture
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The experimental group (Experimental): In this group, the condylar reductor was applied in the surgical treatment of mandibular condylar fractures.
  Interventions: Device: Condylar reductor
- The control group (No Intervention): In this group, traditional surgical instruments were applied in the surgical treatment of mandibular condylar fractures.

INTERVENTIONS:
Device: Condylar reductor — A new surgical instrument was designed to assist the surgeons to perform condylar fracture reduction.
  Arms: The experimental group

SUMMARY:
In condylar fracture surgery, reduction is the most difficult step and the key factor which determined the postoperative outcome. Therefore, the aim of this study is to develop a new instrument, which the investigators call condylar redactor, to assist the surgeon to reduct the condylar segments effectively.

DETAILED DESCRIPTION:
In this prospective cohort study, it involved condylar fractures patients who were received surgical treatment from January 2014 to June 2016. Patients in the experimental group were treated with the condylar reductor, and patients in the control group were treated with the traditional surgical instruments. The primary outcome variable was reduction time and reduction rate. The continuity correction X2 and test student t test were used.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-60 with mandibular condylar fractures were treated in Oral and maxillofacial surgery department, West China hospital of stomatology, China from January 2014 to January 2016.

Exclusion Criteria:

* patients refused to participate in the clinical trial;
* condylar fracture dislocation was not obvious, conservative treatment can be used;
* mandibular condylar comminuted fracture;
* mandibular condyle need to be reconstructed.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
intraoperative reduction time | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Lei Liu, MD, Study Director — West China Hospital of Stomotalogy

REFERENCES:
- See also: The West China Hospital of Stomatology has long been ranked as one of the national top hospitals in China — http://www.hxkq.org/